CLINICAL TRIAL: NCT02504034
Title: Interventional Radiology for the Treatment of Symptomatic Portal Hypertension in Patients With Cavernous Transformation of Portal Vein
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zaibo Jiang, Department of Radiology, The Third Affiliated Hospital, Sun Yat-Sen University, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DORNO3HSYSU
Record Dates: First submitted 2015-07-15; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Portal Vein, Cavernous Transformation Of; Hypertension, Portal
Keywords: Portal Vein, Cavernous Transformation Of; Hypertension, Portal; Radiology, Interventional; Portalsystemic shunt
MeSH Terms: conditions — Portal Vein, Cavernous Transformation Of; Hypertension, Portal

ARMS (1):
- Transhepatic portosystemic shunt (Experimental): Patients with cavernous transformation of portal vein undergo transhepatic portalsystemic shunt and other interventional radiology treatment
  Interventions: Procedure: Transhepatic portosystemic shunt; Device: 6-French sheath; Device: 22-gauge chiba needle; Device: 260-cm-long stiff shaft wire; Device: Balloon catheter; Device: Bare metal stent; Device: Covered stent

INTERVENTIONS:
Procedure: Transhepatic portosystemic shunt — Portal vein (PV) was punctured with a 22-gauge chiba needle. A 0.018-inch guidewire was advanced through the needle into PV lumen. The needle was exchanged and a 6-French sheath inserted over the wire. Then middle hepatic vein (MHV) was punctured with a 20-gauge reformed needle through the transhepatic sheath. Another 0.018-inch guidewire was advanced through the needle into right internal jugular vein and then snared out of body. A 0.035-inch, 260-cm-long stiff shaft wire was introduced through the transjugular sheath and manipulated into main portal vein (MPV) and then into SMV. The parenchymal tract was dilated with balloon catheter, then one or more bare metal stents and one or more covered stents were inserted to line the parenchymal tract.
Device: 6-French sheath
Device: 22-gauge chiba needle
Device: 260-cm-long stiff shaft wire
Device: Balloon catheter
Device: Bare metal stent
Device: Covered stent

SUMMARY:
To evaluate the values of portosystemic shunt and other interventional radiology approaches for treatment of symptomatic portal hypertension in patients with cavernous transformation of portal vein.

ELIGIBILITY:
Inclusion Criteria:

* All patients with portal hypertention who have enough image information to confirm cavernous transformation of portal vein.

Exclusion Criteria:

* Patients with known severe dysfunction of heart, lung, brain, kidney and other vital organs.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-10; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of Gastrointestinal Bleeding | 1 month
  No gastrointestinal bleeding proved by patients' symptoms (If the patients had the history of gastrointestinal bleeding before)
Ascites Volume (mL) | 1 month
  No ascites proved by CT scanning or ultrasound (If the patients had the history of ascites before)

CONTACTS AND LOCATIONS:
Overall Officials: Zaibo Jiang, MD., Study Chair — Sun Yat-sen University
Locations (1):
- Department of Radiology, Guangzhou, Guangdong, China